CLINICAL TRIAL: NCT03211299
Title: Determinants of Liver Fat Composition in Overweight and Obese Humans
Brief Title: Determinants of Liver Fat Composition
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: NL60263.068.16
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Fatty Liver, Nonalcoholic; Insulin Sensitivity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IHL <5%: overweight and obese humans with a liver fat percentage <5%
- IHL 5-10%: overweight and obese humans with a liver fat percentage 5-15%
- IHL >15%: overweight and obese humans with a liver fat percentage >15%

SUMMARY:
Excessive fat in the liver, in absence of high alcohol consumption, is diagnosed as non-alcoholic fatty liver (NAFL). NAFL prevalence is as high as 50-70% in obese people and is associated with impairments in metabolic health, e.g. insulin resistance. Not only the amount, but also the composition of the fat stored in the liver appears to be linked to health outcome measures, such as insulin resistance, but this evidence comes mainly from animal studies. Since fat composition has been linked to health outcome measures, it is important to understand what determines the fatty acid composition of liver fat. De novo lipogenesis (DNL) and adipose tissue fat composition are factors that could determine liver fat composition. Since the end product of DNL are saturated fatty acids and as the majority of fatty acids in the liver originate from adipose tissue, both may influence hepatic fatty acid composition profoundly. Here, our primary hypothesis is that DNL is associated with the relative amount of saturated fatty acids in the liver in overweight/obese humans differing in liver fat content. Furthermore, we hypothesise that adipose tissue fat composition is associated with liver fat composition and that liver fat composition is associated with liver, muscle and whole body insulin sensitivity in overweight/obese humans differing in liver fat content. To this end, liver fat composition, adipose tissue fat composition, DNL and insulin sensitivity will be measured in overweight/obese participants differing in liver content.

DETAILED DESCRIPTION:
Rationale: Excessive fat in the liver, in absence of high alcohol consumption, is diagnosed as nonalcoholic fatty liver (NAFL). NAFL prevalence is as high as 50-70% in obese people and is associated with impairments in metabolic health, e.g. insulin resistance. Not only the amount, but also the composition of the fat stored in the liver appears to be linked to health outcome measures, such as insulin resistance, but this evidence comes mainly from animal studies. Since fat composition has been linked to health outcome measures, it is important to understand what determines the fatty acid composition of liver fat. De novo lipogenesis (DNL) and adipose tissue fat composition are factors that could determine liver fat composition. Since the end product of DNL are saturated fatty acids and as the majority of fatty acids in the liver originate from adipose tissue, both may influence hepatic fatty acid composition profoundly. Up to now, associations between hepatic fatty acid composition, DNL and adipose tissue fatty acid composition have never been determined in the same study.

Objective: The primary objective of this study is to determine the association between DNL and hepatic %SFA in overweight/obese subjects differing in liver fat content. The secondary objectives are to determine the association between adipose tissue fat composition and liver fat composition and to determine the association between liver fat composition and whole body, liver and muscle insulin sensitivity.

Study design: This is a cross-sectional observational study. For this study a design of 3 groups with different amounts of liver fat are included, in order to create a study population with a continuum in liver fat content.

Study population: Twenty-two healthy overweight/obese males and females, aged between 45-70 years and BMI between 27-35 kg/m2 will participate in the whole study. To create a continuum in liver fat content, eight subjects with liver fat content lower than 5% and 14 subjects with liver fat content higher than 5%, of which at least seven subjects have a liver fat content of at least 15%, will be included. To be able to include enough people in each group, around 31 participants will be included in total. A part of the participants will stop participating in the study after determination of liver fat content (in case the liver fat content does not match the groups).

Main study parameters/endpoints: The primary study parameters are %SFA in the liver and DNL. %SFA in the liver will be determined using MRS and DNL will be determined by applying stable isotope techniques. The secondary study parameters are hepatic fat composition, measured as %MUFA and %PUFA in addition to %SFA using MRS, adipose tissue fat composition, determined using MRS and biopsies, and insulin sensitivity, measured by a hyperinsulinemic euglycemic 2- step clamp.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Caucasian (people will be excluded when having a 50% or a more then 50% racial African/Asian background)
* Male or postmenopausal female
* Aged 45-70 years at start of the study
* Body mass index (BMI) 27 - 35 kg/m2
* Stable dietary habits (no weight loss or gain >3kg in the past 3 months)
* Sedentary lifestyle (not more than 2 hours of sports per week)

Exclusion Criteria:

* Type 2 diabetes
* Active diseases (cardiovascular, diabetes, liver, kidney, cancer or other)
* Contra-indication for MRI (which can be found in appendix I)
* Alcohol consumption of >2 servings per day
* Smoking >5 cigarettes per day
* Use of anti-coagulants

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty-two healthy overweight/obese males and females, aged between 45-70 years and BMI between 27-35 kg/m2 will participate in the whole study. To create a continuum in liver fat content, eight subjects with liver fat content lower than 5% and 14 subjects with liver fat content higher than 5% (NAFL) will be included. At least seven volunteers with NAFL will have severely elevated hepatic fat content (liver fat percentage ≥ 15%).
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
%SFA in the liver | 20 minutes
  expressed as relative amount of SFA to the total amount of fatty acids (determined by magnetic resonance spectroscopy)
DNL | 16 hours
  expressed as percentage of palmitate in VLDL-TG originating from DNL (determined by use of deuterium water)

SECONDARY OUTCOMES:
Liver fat composition | 20 minutes
  expressed as relative amount of MUFA and PUFA to the total amount of fatty acids, in addition to %SFA (determined by magnetic resonance spectroscopy)
Adipose tissue fat composition | 20 minutes
  expressed as relative amount of SFA, MUFA and PUFA to the total amount of fatty acids (determined by magnetic resonance spectroscopy and from subcutaneous adipose tissue biopsy)
Adipose tissue fat composition | 15 minutes
  expressed as relative amount of linoleic acid, docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA) to the total amount of fatty acids (determined from subcutaneous adipose tissue biopsy)
Hepatic insulin sensitivity | 8.5 hours
  expressed as % suppression of endogenous glucose production (EGP)(determined by hyperinsulinemic euglycemic clamp).
Muscle insulin sensitivity | 15 minutes
  expressed as determinants/markers for muscle insulin sensitivity in muscle biopsy (oxphos, GLUT4, intramyocellular lipids (IMCL).
peripheral insulin sensitivity | 8.5 hours
  expressed as rate of disappearance (Rd) in μmol/kg/min (determined by hyperinsulinemic euglycemic clamp).
whole body insulin sensitivity | 8.5 hours
  expressed as glucose infusion rate (GIR) in μmol/kg/min (determined by hyperinsulinemic euglycemic clamp).

OTHER OUTCOMES:
Intrahepatic fat accumulation | 10 minutes
  expressed as % (determined by magnetic resonance spectroscopy)
body composition | 15 minutes
  expressed as fat mass (%) and fat-free mass (%) (determined by BodPod)
abdominal visceral adipose tissue and abdominal subcutaneous adipose tissue | 10 minutes
  expressed as % (determined by magnetic resonance spectroscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Vera B Schrauwen, Dr, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Roumans KHM, Lindeboom L, Veeraiah P, Remie CME, Phielix E, Havekes B, Bruls YMH, Brouwers MCGJ, Stahlman M, Alssema M, Peters HPF, de Mutsert R, Staels B, Taskinen MR, Boren J, Schrauwen P, Schrauwen-Hinderling VB. Hepatic saturated fatty acid fraction is associated with de novo lipogenesis and hepatic insulin resistance. Nat Commun. 2020 Apr 20;11(1):1891. doi: 10.1038/s41467-020-15684-0. PMID 32312974